CLINICAL TRIAL: NCT02517606
Title: Hip Posterolateral Complex Strengthening in Patients With Chronic Nonspecific Low Back Pain: a Randomized Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Bahia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado da Bahia (Other)
Responsible Party: Principal Investigator, Mansueto Gomes Neto, Dr Mansueto Gomes Neto, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUBahia LBP
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional physical therapy plus HPCS (Experimental): Conventional physical therapy (Combination of manual therapy techniques and exercises for spinal segmental stabilization) plus the addition of hip posterolateral complex strengthening (HPCS)
  Interventions: Other: Conventional physical therapy plus HPCS
- Conventional physical therapy (Active Comparator): Conventional physical therapy (Combination of manual therapy techniques and exercises for spinal segmental stabilization)
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Conventional physical therapy plus HPCS — Conventional physical therapy plus the addition of hip posterolateral complex strengthening
  Arms: Conventional physical therapy plus HPCS
Other: Conventional physical therapy — Conventional physical therapy (combination of manual therapy techniques and exercises for spinal segmental stabilization)
  Arms: Conventional physical therapy

SUMMARY:
Chronic nonspecific low back pain is an important health condition with a high prevalence worldwide and it is associated with enormous direct and indirect costs to the society. Clinical practice guidelines show that many interventions are available to treat patients with chronic low back pain, but the vast majority of these interventions have a modest effect in reducing pain and disability. A biomechanical approach that has been raised is that a weakness of the hip abductors, extensors, and lateral rotators musculature (posterolateral complex - PLC) would lead to excessive contralateral pelvic drop during weight-bearing activities such as walking, running, climbing up or downstairs, generating an overload in the lumbar area. Although the strengthening of the hip PLC is largely used in clinical practice for treating patients with hip and knee injuries, there is still a lack of evidence regarding patients with low back pain. Therefore, questions remain about the efficacy of the hip dynamic stabilization as an additional intervention to conventional treatment in a well design trial with statistic power.

DETAILED DESCRIPTION:
Randomised clinical trial will be held in following the recommendations of the CONSORT (Consolidated Standards of Reporting Trials). Will be recruited participants of both genders, aged between 18 and 60 years, with and without chronic nonspecific low back pain for over 3 months without irradiation for lower limbs. Potential participants with chronic nonspecific low back pain will be referred by their doctors orthopedic surgeons and/or rheumatologists that will make all the assessments and routine exams, for example, Imaging tests, prescription drugs and referral to physical therapy care. The characteristics of participants will be collected through an evaluation form specially designed for this study. This assessment form will contain issues related to demographic and anthropometric data, plus information about the clinical picture of the participants, as for example the use of medications, physical activity level, educational level, prior history of back pain and duration of symptoms.The clinical outcomes will be obtained at the completion of treatment (6 weeks) and at 3, 6, and 12 months after randomization.

The data will be collected by a blinded assessor. The statistical analysis will follow the intention-to-treat principles.

ELIGIBILITY:
Inclusion Criteria:

* • Will be included 70 patients of both sexes, adults with medical diagnosis divided into two groups: Group A consisted of 35 patients use receive conventional physical therapy plus the addition of hip PLC strengthening and group B consisted of 35 patients also only use conventional physical therapy

Exclusion Criteria:

* Will be excluded from the study patients who have neurological or osteoarticular disease preventing the ambulation of these individuals.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 weeks
  The numerical visual scale evaluates levels of intensity of pain perceived by the patient through a range of 11 points (ranging from 0 to 10), 0 being no pain and 10 rank as the worst pain possible. Participants will be instructed to report the level of pain intensity based on the last 7 days.
Disability | 6 weeks
  The Roland Morris disability questionnaire is an instrument widely used in research and clinical practice for evaluation of functional disability associated with back pain through 24 issues that describe everyday situations in which patients have difficulty to carry out due low back pain.

SECONDARY OUTCOMES:
Strength | 6 weeks
  A previously calibrated manual hand-held dynamometer will be used to measure maximum isometric strength of abduction and hip extension
Functioning (activities and participation) | 6 weeks
  The World Health Organization Disabilty Assessment Schedule (WHODAS 2.0) 2.0 is a tool developed by the World Health Organization (who) to assess the limitations in activities and participation restrictions already adapted and validated in Brazil. The WHODAS 2.0 was designed to evaluate the functionality in 6 areas of activity: cognition, mobility, self-care, interpersonal relationships, daily activities and Participation.
Movement analysis with a 2-D system | 6 weeks
  The gait and step down kinematic parameters will be calculated with SIMI Reality Motion Systems. The subjects will be fitted with colors markers on the lower limbs and trunk. Our approach automatically processes video sequences gathered with a digital camera and extract the 2D joints' location and their angle trend over time. The peaks of the movements of the hip, pelvis and trunk in the frontal and sagittal planes will be evaluated and compared between groups before and after treatment.

OTHER OUTCOMES:
Pain | 6 months
  The numerical visual scale evaluates levels of intensity of pain perceived by the patient through a range of 11 points (ranging from 0 to 10), 0 being no pain and 10 rank as the worst pain possible. Participants will be instructed to report the level of pain intensity based on the last 7 days.
Disability | 6 months
  The Roland Morris disability questionnaire is an instrument widely used in research and clinical practice for evaluation of functional disability associated with back pain through 24 issues that describe everyday situations in which patients have difficulty to carry out due low back pain.
Functioning (activities and participation) | 6 months
  The World Health Organization Disabilty Assessment Schedule (WHODAS 2.0) 2.0 is a tool developed by the World Health Organization (who) to assess the limitations in activities and participation restrictions already adapted and validated in Brazil. The WHODAS 2.0 was designed to evaluate the functionality in 6 areas of activity: cognition, mobility, self-care, interpersonal relationships, daily activities and Participation.

CONTACTS AND LOCATIONS:
Overall Officials: Mansueto G Neto, Principal Investigator — UFBA
Locations (1):
- Mansueto Gomes Neto, Salvador, Estado de Bahia, Brazil